CLINICAL TRIAL: NCT04331717
Title: BASH-PC: Bariatric Arterial Embolization for Men Starting Hormones for Prostate Cancer
Brief Title: Bariatric Arterial Embolization for Men Starting Hormones for Prostate Cancer
Acronym: BASH-PC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: accrual on hold
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Maryland Cigarette Restitution Fund (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: J1943; IRB00207275 (Other: JHM IRB)
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Prostate Adenocarcinoma; Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Diet and exercise with BAE (Experimental): After enrollment in the clinical trial, all men will be enrolled in diet and exercise counseling through the weight management program for a total of 4 weeks. If participants lose >5 pounds of total body weight from weight management alone in the first 4 weeks, these participants will be excluded from study and will not undergo BAE but will be encouraged to continue with weight management. Those still enrolled will undergo BAE. Within 7 days of BAE, men will be given ADT (lupron subcutaneous injection).
  Interventions: Device: Bead Block 300-500 um; Behavioral: Weight Management; Drug: Lupron

INTERVENTIONS:
Device: Bead Block 300-500 um — These patients will undergo embolization with 300-500µm Bead Block particles.
Behavioral: Weight Management — All participants will be enrolled in weight management through the Johns Hopkins Weight Management Center. During weeks -4 through 0, participants will be required to go to weekly visits. Weight management will include counseling on diet, exercise and behavior change. Food programs, pharmacotherapy and other procedures will not be utilized.
Drug: Lupron — 22.5 mg will be given as a single intramuscular or subcutaneous injection once every 12 weeks according to the standard of care for prostate cancer. If leuprolide acetate, 22.5 mg for 3-month administration is not available, a suitable substitute may be allowed upon approval by the principle investigator

SUMMARY:
The standard of care for obese men starting Androgen deprivation therapy (ADT) is physician based dietary and exercise counseling. Interventions to lessen the harmful effects of ADT are needed yet have been limited. Exercise is one strategy that has been attempted however there is conflicting data as to whether or not exercise effectively improves body mass, results in sustained weight loss, improvements in metabolic risk profiles including glucose tolerance and lipid profiles in men starting ADT, or has any effect of progression of cancer. Dietary interventions have been attempted without clear improvement in weight, metabolic factors, quality of life or cancer progression. Bariatric arterial embolization (BAE), given it results in weight loss in obese men and women without cancer, may be able to stave off the harmful side effects of ADT by inducing weight loss. Therefore, the investigators hypothesize that Bariatric Arterial embolization (BAE), done prior to initiation of ADT, will mitigate the weight gain and metabolic side effects associated with ADT, by inducing weight loss of at least 5% in obese men with biochemical recurrent prostate cancer starting ADT.

The primary objective is to determine if BAE, done prior to ADT initiation in obese men (with obesity related comorbid condition) with biochemically recurrent prostate cancer, can induce 5% or greater weight loss at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information (HIPAA authorization will be included in the informed consent)
* Males aged 18 years of age and above
* Histological proof of adenocarcinoma of the prostate
* Non-metastatic disease by computed tomography (CT), magnetic resonance imaging (MRI) or Nuclear medicine (NM) bone scan. Patients must have CT abdomen/pelvis with contrast prior to enrollment.
* Metastatic disease may be permitted if NOT starting on any concomitant therapy (ie chemotherapy, anti-androgens)
* Prior local therapy with prostatectomy or radiotherapy (including brachytherapy) or both
* BMI >30 kg/m2 with a concurrent obesity related comorbidity

Obesity related comorbidity is defined as:

* hypertension (resting blood pressure >130/80 millimeters of mercury (mmHg) or being on medication to treat high blood pressure50),
* coronary artery disease (defined as prior myocardial infarction, elevated coronary artery calcium score, positive stress test history),
* dyslipidemia (triglyceride level of >150mg/dL or being on medicine to treat high triglycerides; HDL < 40mg/dL or being on medicine to treat cholesterol)51,
* diabetes (fasting glucose >126mg/dL, A1c > 6.5% or on medication for diabetes)52,
* pre-diabetes (fasting plasma glucose 100-125mg/dL)52,
* elevated waist circumference (>40 inches in men),
* obstructive sleep apnea,
* arthritis, or
* non-alcoholic steatohepatitis.
* Prior salvage or adjuvant radiation therapy is allowed but must have been completed at least 3 months prior to enrollment
* Non-castrate levels of testosterone (>50 ng/dL required)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening
* Vascular anatomy (including celiac, hepatic and gastric arteries) that in the opinion of the interventional radiologist is amenable to bariatric embolization as assessed on 3D CT angiography
* Participants must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days Absolute neutrophil count (ANC) ≥ 1.0 x 109/L Platelet count ≥ 50 x 109/L Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) < 2.5 x institutional upper limit of normal Estimated Glomerular filtration rate (GFR) >60ml/min

Exclusion Criteria:

* Prior hormonal therapy within 12 months of enrollment
* Planned concurrent cytotoxic chemotherapy or antiandrogens (ex. bicalutamide, abiraterone acetate, enzalutamide or any investigational agent).
* Contraindication to the use of leuprolide, such as a previous hypersensitivity reaction to an Luteinizing hormone-releasing hormone (LHRH) analogue or any of the excipients in the leuprolide injection
* Prior history of gastric, pancreatic, hepatic and/or splenic surgery
* Prior radiation therapy to the upper abdomen (pelvic radiation is not an exclusion)
* Prior embolization to the stomach, spleen or liver
* Cirrhosis or known portal venous hypertension
* Active peptic ulcer disease or significant risk factors for peptic ulcer disease including daily NSAID use or daily smoking
* Hiatal hernia >5cm in size
* Active h.pylori infection (patients will be required to have negative h.pylori testing)
* Weight >400 pounds or BMI >45kg/m2
* Known aortic arch pathology such as aneurysm or dissection
* Major comorbidity that precludes procedure including significant cardiovascular disease or peripheral arterial disease including the following:

Myocardial infarction within 6 months before screening Unstable angina within 3 months before screening New York Heart Association class III or IV congestive heart failure or a history of New York Heart Association class III or IV congestive heart failure unless a screening echocardiogram or multi-gated acquisition scan performed within 3 months before the randomization date demonstrates a left ventricular ejection fraction ≥ 45% History of clinically significant ventricular arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes) Uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure measurements showing systolic blood pressure > 170 mm Hg or diastolic blood pressure > 105 mm Hg at screening Peripheral arterial stenting or bypass procedure within 6 months before screening Active claudication

* Diabetes with A1c >7% or requiring medication other than metformin
* Known gastric motility dysfunction
* Preexisting chronic abdominal pain
* Positive stool occult study
* Inflammatory bowel disease
* Known history of allergy to iodinated contrast media
* American Society of Anesthesiology (ASA) physical status classification system Class 4 of 5 (very high risk surgical candidates: class 4 = incapacitating disease that is a constant threat to life) at the time of screening for enrollment
* Any condition in which the principle investigator feels participation in the trial would put the patient and undue risk

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience at least 5 percent weight loss | At 6 months
  Number of participants who experience at least 5 percent weight loss at 6 months after BAE.

SECONDARY OUTCOMES:
Number of adverse events | Up to 6 months
  Number of adverse events will be assessed to determine if there are any increased adverse events in men with prostate cancer undergoing BAE.
Change in Blood Pressure | Baseline, weeks 4, 8, 12, 16, 20, 24, 36 and 48
  Blood pressure (mmHg) will be assessed for changes over the specified time points.
Change in Respiratory Rate | Baseline, weeks 4, 8, 12, 16, 20, 24, 36 and 48
  Respiratory rate in breaths per minute will be assessed for changes over the specified time points.
Change in Oxygen saturation | Baseline, weeks 4, 8, 12, 16, 20, 24, 36 and 48
  Oxygen saturation (percentage) will be assessed for changes over the specified time points.

OTHER OUTCOMES:
Time to disease progression | Up to 51 weeks
  The amount of Time (months) till prostate-specific antigen (PSA) progression which will be assessed by PSA blood test at screening, 12 weeks, 24 weeks, 36 weeks, and 48 weeks. With PSA progression defined as first PSA increase that is 25% and 2ng/mL above the nadir, and which is confirmed by a second value at least 3 weeks later, or the amount of Time till radiographic progression which will be assessed by RECIST v1.1 using conventional CT chest/abd/pelvis or NM Bone scan. Radiographic progression will be defined as visceral and nodal disease or at least 2 new bone lesions.
Change in C-Reactive Protein level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  C-Reactive Protein (CRP) levels in mg/dL.
Change in Erythrocyte Sedimentation Rate | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Erythrocyte Sedimentation Rate (ESR) in millimeters per hour.
Change in Interleukin 6 level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Interleukin 6 (IL-6) levels in pg/ml.
Change in Interleukin 8 level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Interleukin 8 (IL-8) levels in pg/mL.
Change in Tumor Necrosis Factor Alpha level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Tumor Necrosis Factor Alpha (TNF-α) levels in pg/mL.
Change in Interleukin 1 alpha level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Interleukin 1 alpha (IL-1α) levels in pg/mL.
Change in Interleukin 1 beta level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Interleukin 1 beta (IL-1β) levels in pg/mL.
Change in Ghrelin level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Ghrelin levels in pg/mL.
Change in leptin level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Leptin levels in percentage.
Change in active Glucagon-like Peptide-1 level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Active Glucagon-like Peptide-1 (GLP-1) levels in pmol/L.
Change in Peptide YY level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Peptide YY (PYY) levels in pmol/L.
Change in Insulin-like growth factor 1 level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Insulin-like growth factor 1 (IGF-1) levels in ng/mL.
Change in Adiponectin level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Adiponectin levels in mL.
Change in microbiome | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  To evaluate changes in the microbiome of men with prostate cancer before and after undergoing BAE and starting ADT.
Change in high density lipoprotein level | At 12 weeks, 24 weeks, 36 weeks and 48 weeks
  High density lipoprotein (HDL) levels in mg/dL.
Change in triglycerides level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Triglycerides level in mg/dL.
Change in fasting glucose level | At 12 weeks, 24 weeks, 36 weeks and 48 weeks
  Fasting glucose (mg/dL) will be assessed at specified time points for any changes. Fasting glucose within normal is <126 mg/dL.
Change in hemoglobin A1c level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Hemoglobin A1c levels in percentage will be assessed at 12 weeks, 24 weeks, 36 weeks, and 48 weeks.
Change in low density lipoprotein level | At 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Low density lipoprotein (LDL) levels in mg/dL.
Change in Quality of life as assessed by Abbreviated version of the medical outcomes, short-form 36 (SF-12) | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Quality of Life scored on a scale from 0 to 48, higher scores representing highest level of functioning possible.
Change in Quality of life as assessed by Impact of Weight on Quality of Life Questionnaire (IWQOL) | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Impact of Weight on Quality of Life all 31 questions are scored on a scale from 1 to 5, higher scores representing poorer quality of life.
Change in Sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  The global PSQI score is calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Change in Quality of life as assessed by Expanded Prostate Cancer Index Composite-26 question assessment (EPIC-26) | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  All questions are scored on a scale from 0 to 100. The total score from all of the questions answered is divided by the total number of the questions answered yielding a global score from 0-100 with 100 representing the highest level of functioning possible.
Change in Fatigue as assessed by the Brief Fatigue Inventory (BFI) | Baseline, 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Fatigue Rated by 9 each item on a 0-10 and 1 on a yes no scale, higher scores representing more fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Marshall, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States